CLINICAL TRIAL: NCT03281057
Title: Community Reinforcement and Family Training (CRAFT)
Acronym: CRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kjeld Andersen (Other)
Responsible Party: Sponsor-Investigator, Kjeld Andersen, Professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRAFT112018
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: CRAFT; Concern Significant Others; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Cluster randomization Clinical trial with 3 arms - individual, group, and self-help intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual CRAFT (Experimental): Individual CRAFT is offered to 135 participants and each participants are going to get 6 sessions.
  Interventions: Behavioral: CRAFT
- Group CRAFT (Experimental): Open group CRAFT is offered to 135 participants in 6 sessions.
  Interventions: Behavioral: CRAFT
- Self-help materials (Experimental): Self-help materials (control group) are going to be offered a self-help book, because it is unethically not to offer any intervention, as the CRAFT intervention in early studies have shown to be very effectful
  Interventions: Behavioral: CRAFT

INTERVENTIONS:
Behavioral: CRAFT — CRAFT is a counseling/therapist to concern significant others to get their loved one, with an alcohol use disorder, into treatment

SUMMARY:
The present study is dedicated to empowering individuals close to an addicted person (i.e. concerned significant others, CSOs) to create changes in their family environment: changes that increase the likelihood of the addicted person seeking treatment.

The Danish National Clinical Guideline for the treatment of alcohol dependence recommends that alcohol treatment centers offer interventions aimed at CSOs, providing them with the support and empowerment that will enable them to motivate the problem drinker to enter treatment. In the US, the Community Reinforcement and Family Training (CRAFT) intervention has been shown to offer the most effective support to CSOs. CRAFT has consistently demonstrated a two to three times' higher impact on getting individual with an alcohol use disorder (AUD) to attend treatment, compared to other kinds of interventions. Studies of the intervention so far have, however, been small, and the format used in the delivery of CRAFT has not been fully investigated.

The aim of the present cluster randomized controlled trial is to implement and investigate CRAFT in a Danish context and with sufficient sample size. Consecutive CSOs will through cluster randomization be randomized to receive either CRAFT in a group format, CRAFT in an individual format, or a control condition, consisting of self-help material only. The primary outcome of the study will be the rate of individuals with AUD entering treatment following the intervention targeted at the CSOs within three months from its initiation. Data will be collected from all CSOs at baseline, three, and six months after baseline.

ELIGIBILITY:
Inclusion criteria:

* 18 years and older
* Being a CSO to a person with AUD who is not currently in treatment for alcohol problems
* Having the intention to maintain the contact during the next 90 days
* Having had regular contact with the problem drinker for the last 90 days (face-to-face contact for several hours on at least a weekly basis) and having the intention to maintain the contact during the next 90 days.
* Being prepared support the problem drinker if he/she chooses to seek treatment, at least to some extent.

Exclusion Criteria:

* Suffering from dementia or other cognitive disorders
* Not speaking Danish
* Being psychotic or otherwise severely mentally ill
* Suffering from AUD in the last three months
* Being concerned about a person who, according to the CSO, mainly use illegal substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Whether the drinker has sought treatment for her/his alcohol use disorder | 3 months after baseline
  The proportion of problem drinkers, who enter alcohol treatment centers from baseline and until three months after their CSOs enrolled in the CRAFT study.

SECONDARY OUTCOMES:
Changes in the anxiety, - depression and concern symptoms of concern significant others following CRAFT intervention | 3 and 6 months after baseline
Improvement in the relationship between the concern significant other and the drinker before and after CRAFT intervention | 3 and 6 months after baseline
  Measured by the Relationship Happiness Scale
Changes in number of sick leave days for concern significant others from 6 months before to 6 months after enrollment in the study. | 6 months after baseline
Changes in quality of life among concern significant others. | 3 and 6 months after baseline
  Measured by WHO's quality of life scale "WHOQol-Bref - Danish version"

CONTACTS AND LOCATIONS:
Overall Officials: Anette Søgaard Nielsen, Ass. Prof., Study Chair — Unit of Clinical Research, University of Southern Denmark
Locations (2):
- Denmark (2):
  - Unit if Clinical Alcohol Research, Odense
  - Research Unit of Psychiatry, Psychiatric Unit Odense - University function, Odense C

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hellum R, Bilberg R, Andersen K, Bischof G, Hesse M, Nielsen AS. Primary Outcome from a cluster-randomized trial of three formats for delivering Community Reinforcement and Family Training (CRAFT) to the significant others of problem drinkers. BMC Public Health. 2022 May 10;22(1):928. doi: 10.1186/s12889-022-13293-8. PMID 35538465
- [Derived] Hellum R, Nielsen AS, Bischof G, Andersen K, Hesse M, Ekstrom CT, Bilberg R. Community reinforcement and family training (CRAFT) - design of a cluster randomized controlled trial comparing individual, group and self-help interventions. BMC Public Health. 2019 Mar 14;19(1):307. doi: 10.1186/s12889-019-6632-5. PMID 30871596